CLINICAL TRIAL: NCT02604615
Title: Two Cycles Versus Four Cycles of Capecitabine Combined Oxaliplatin Concurrent Radiotherapy as First-line Therapy for Chinese Locally Advanced Esophageal Squamous Cell Carcinomas, an Open Randomised Phase III Cilinical Trial
Brief Title: The Role of Different Cycles of Chemotherapy（Capecitabine-oxaliplatin） in Esophageal Chemoradiotherapy
Acronym: DCOECRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Xinyang Central Hospital (Other); Anyang Tumor Hospital (Other); No. 150 Central Hospital of the Chinese People Liberation Army (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: capecitabine-oxaliplatin
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms
Keywords: Chemoradiotherapy; Esophageal Squamous Cancer; Capecitabine and oxaliplatin; Chinese; Randomized Controlled Trials
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine-oxaliplatin 2 cycles (Experimental): oxaliplatin：65mg/m2,d1,8,22,29,I.V; capecitabine: 625mg/m2, bid d1-5; q1w, po,5 weeks in total; radiotherapy:50Gy,2 Gy/d,5d/w.
  Interventions: Drug: Capecitabine(Aibin); Drug: Oxaliplatin(Aiheng); Radiation: Radiotherapy
- Capecitabine-oxaliplatin 4 cycles (Active Comparator): oxaliplatin:65mg/m2,d1,8,22, 29,43,50,64,71,I.V; capecitabine:625mg/m2,bid d1-5; q1w, po,10 weeks in total; radiotherapy:50Gy ,2 Gy/d,5d/w.
  Interventions: Drug: Capecitabine(Aibin); Drug: Oxaliplatin(Aiheng); Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine(Aibin) — capecitabine(Aibin):625mg/m2,bid d1-5; q1w, po,5 or 10 weeks in total
  Other Names: Aibin
Drug: Oxaliplatin(Aiheng) — Oxaliplatin(Aiheng):65mg/m2,d1,8,22,29,I.V. or Oxaliplatin(Aiheng):65mg/m2,d1,8,22,29,43,50,64,71,I.V.
  Other Names: Aiheng
Radiation: Radiotherapy — concurrent radiotherapy:50Gy in total,2 Gy/d,5d/w,Until disease progression or unacceptable toxicity
  Other Names: Radiation Therapy

SUMMARY:
A two-arm (two cycles' versus four cycles' capecitabine combined oxaliplatin concurrent radiotherapy) randomised Phase III clinical trial was started in Oct. 2015. Definitive chemoradiotherapy is the standard regimen in Western countries for patients with esophageal cancer who can't receive surgery or reject surgery. But in China because of its severer toxic reaction, most of patients had to discontinue treatment at the halfway way. Thus, the chemotherapy regimen of capecitabine combined oxaliplatin are widely used in clinical due to its characristic of low toxic reaction.

The purpose of this study is to confirm the efficacy and safety of the different cycles(two cycles and four cycles ) of Capecitabine-oxaliplatin in Chinese esophageal squamous carcinoma radical concurrent chemoradiotherapy. A total of 60 patients will be accrued from China within 2 years. The primary endpoint is overall survival and the secondary endpoints include progression-free survival, response rate, pathologic complete response rate and adverse events.

DETAILED DESCRIPTION:
First: The investigators use excel generate a 5 digits random number table. After subjects sign the informed consent, investigators will chose one for themm. Subject who get an odd number will receive 2cycles' chemotheapy concurrent radiotherapy and even number receive 4cycles'. Investigators should record the congruent relationship of subjects with group code.

Second: The investigators are required to record subjects' base measurements. The base measurements items:1.Tumor confirmed date,TNM staging,History of esophageal cancer treatment;2.Demographic data,past medical history;3.physical examination(a detailed system check including general neurological examination);4.vital signs,Height,Weight;5.PS score,Quality of life;6.serum biochemistry(ALT,AST,AKP,TBIL,blood glucose,BUN,Ccr,electrolyte,et al.);7. Blood RT(RBC,HGB,WBC,ANC,PLT,et al.);8.Urine routines;9.Endoscopic biopsy(More than 3 pieces of biopsy specimens),chest CT,abdomen ultrasound/CT/MRI,PET-CT,et al.;10.Blood/urine pregnancy tests;11.Collect blood samples(5 ml);12.Preserve CorpseSample. note:Check the time limit-2 weeks before get into groups.

Third:Observation items during treatment include 3-8 items of the base measurements;Radiotherapy 20 times, should review of esophageal barium meal or chest CT. The investigators need to observe adverse event during treatment and eveluate the relationship of adverse event with researched therapeutic regimen according to the Common Terminology Criteria for Adverse Events,CTCAE) (V4.0, 2009-05-28) and accurately fill in Case Report Form(CRF).

Fourth: Follow-up items include 3-9 items of the base measurements;bood and tissue sample should also be preserved when subject receives 16th weeks' review.

The patient who withdrew from the study during researched treatment must accept the end evaluation research. The investigators must record the reason and the date of termination in patient' progress note and CRF.

Cases of complete report should transfer to data administrators after investigates by clinical research associate. Data administrators input and management data.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and signed a consent form
* Histologically proven squamous cell carcinoma of the esophagus, initial treatment (Not had surgery, radiotherapy, chemotherapy or targeted therapy)
* the tumor was in T2-4N0-2M0, locally advanced（AJCC2002）
* Have a measurable lesions.
* Male or female who has fertility is willing to take contraceptive measures in the experiment
* WBC≥3x10 9/L；Hb≥80g/L；ANC ≥1.5x10 9/L；PLT ≥100x10 9/L；TBIL< 1.5xN；AST (SGOT)/ALT (SGPT) ≤2.5xN；Cr≤1.5xN.
* Performance status score 0-2
* Expected lifetime>3 months

Exclusion Criteria:

* Pregnant, lactating women or With fertility but did not use contraceptive measures
* Has a history of severe allergic or idiosyncrasy
* Hab been treated with surgery, radiation and chemotherapy or targeted therapy for esophageal cancer
* After exploratory thoracotomy or Laying an esophageal tracheal stent
* Received a major surgery treatment within 28 days prior to the start of research and treatment
* History of organ transplantation
* Has uncontrolled seizures or Lose self-knowledge because of mental illness
* Severe infection
* Oral capecitabine who have difficulty with,such as esophageal obstructed completely, dysphagia,The activities of digestive ulcer, Gastrointestinal bleeding
* Severe chronic diseases, such as, hepatopathy, nephropathy, respiratory disease,high blood pressure, diabetes.
* Other malignant tumor in recent 5 years.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
overall survival, OS | 2 years

SECONDARY OUTCOMES:
progression-free survival,PFS | 2 years
overall remission rate, ORR | 16 weeks
serious adverse event，SAE | 16 weeks
quality of life, Qol | 16 weeks
pathologic complete response rate | 16 weeks
disease control rate,DCR | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology; Tanyou Shan, Master, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Xiaoshan Feng, Doctor, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Jiachun Sun, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xinshuai Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Guoqiang Kong, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Xiaozhi Yuan, Master, Study Director — The First Affiliated Hospital of Henan University of Science and Technology; Ruinuo Jia, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Zhou, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Jing Ren, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Ruina Yang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Dan Wang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yongxuan Liu, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Yali Zhang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Weijiao Yin, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Wei Wang, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology; Shiyuan Song, Master, Principal Investigator — The First Affiliated Hospital of Henan University of Science and Technology
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Park JW, Kim JH, Choi EK, Lee SW, Yoon SM, Song SY, Lee YS, Kim SB, Park SI, Ahn SD. Prognosis of esophageal cancer patients with pathologic complete response after preoperative concurrent chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):691-7. doi: 10.1016/j.ijrobp.2010.06.041. Epub 2010 Oct 1. PMID 20888705
- [Background] Fakhrian K, Ordu AD, Haller B, Theisen J, Lordick F, Bisof V, Molls M, Geinitz H. Cisplatin- vs. oxaliplatin-based radiosensitizing chemotherapy for squamous cell carcinoma of the esophagus: a comparison of two preoperative radiochemotherapy regimens. Strahlenther Onkol. 2014 Oct;190(11):987-92. doi: 10.1007/s00066-014-0661-x. Epub 2014 Apr 16. PMID 24737541
- [Background] Pera M, Gallego R, Montagut C, Martin-Richard M, Iglesias M, Conill C, Reig A, Balague C, Petriz L, Momblan D, Bellmunt J, Maurel J. Phase II trial of preoperative chemoradiotherapy with oxaliplatin, cisplatin, and 5-FU in locally advanced esophageal and gastric cancer. Ann Oncol. 2012 Mar;23(3):664-670. doi: 10.1093/annonc/mdr291. Epub 2011 Jun 7. PMID 21652581
- [Background] Qin TJ, An GL, Zhao XH, Tian F, Li XH, Lian JW, Pan BR, Gu SZ. Combined treatment of oxaliplatin and capecitabine in patients with metastatic esophageal squamous cell cancer. World J Gastroenterol. 2009 Feb 21;15(7):871-6. doi: 10.3748/wjg.15.871. PMID 19230050
- [Background] Chiarion-Sileni V, Innocente R, Cavina R, Ruol A, Corti L, Pigozzo J, Del Bianco P, Fumagalli U, Santoro A, Ancona E. Multi-center phase II trial of chemo-radiotherapy with 5-fluorouracil, leucovorin and oxaliplatin in locally advanced esophageal cancer. Cancer Chemother Pharmacol. 2009 May;63(6):1111-9. doi: 10.1007/s00280-008-0834-3. Epub 2008 Sep 30. PMID 18825381
- [Background] O'Connor BM, Chadha MK, Pande A, Lombardo JC, Nwogu CE, Nava HR, Yang G, Javle MM. Concurrent oxaliplatin, 5-fluorouracil, and radiotherapy in the treatment of locally advanced esophageal carcinoma. Cancer J. 2007 Mar-Apr;13(2):119-24. doi: 10.1097/PPO.0b013e318046ee1a. PMID 17476140
- [Background] Lee SJ, Kim S, Kim M, Lee J, Park YH, Im YH, Park SH. Capecitabine in combination with either cisplatin or weekly paclitaxel as a first-line treatment for metastatic esophageal squamous cell carcinoma: a randomized phase II study. BMC Cancer. 2015 Oct 14;15:693. doi: 10.1186/s12885-015-1716-9. PMID 26468007
- [Background] Xing L, Liang Y, Zhang J, Wu P, Xu D, Liu F, Yu X, Jiang Z, Song X, Zang Q, Wang W. Definitive chemoradiotherapy with capecitabine and cisplatin for elder patients with locally advanced squamous cell esophageal cancer. J Cancer Res Clin Oncol. 2014 May;140(5):867-72. doi: 10.1007/s00432-014-1615-5. Epub 2014 Mar 1. PMID 24578238
- [Background] Koo DH, Park SI, Kim YH, Kim JH, Jung HY, Lee GH, Choi KD, Song HJ, Song HY, Shin JH, Cho KJ, Yoon DH, Kim SB. Phase II study of use of a single cycle of induction chemotherapy and concurrent chemoradiotherapy containing capecitabine/cisplatin followed by surgery for patients with resectable esophageal squamous cell carcinoma: long-term follow-up data. Cancer Chemother Pharmacol. 2012 Mar;69(3):655-63. doi: 10.1007/s00280-011-1750-5. Epub 2011 Oct 4. PMID 21968953
- [Background] Lee SJ, Ahn BM, Kim JG, Sohn SK, Chae YS, Moon JH, Lee EB, Kim JC, Park IK, Jeon SW. Definitive chemoradiotherapy with capecitabine and cisplatin in patients with esophageal cancer: a pilot study. J Korean Med Sci. 2009 Feb;24(1):120-5. doi: 10.3346/jkms.2009.24.1.120. Epub 2009 Feb 28. PMID 19270824
- [Background] Lee J, Im YH, Cho EY, Hong YS, Lee HR, Kim HS, Kim MJ, Kim K, Kang WK, Park K, Shim YM. A phase II study of capecitabine and cisplatin (XP) as first-line chemotherapy in patients with advanced esophageal squamous cell carcinoma. Cancer Chemother Pharmacol. 2008 Jun;62(1):77-84. doi: 10.1007/s00280-007-0577-6. Epub 2007 Aug 31. PMID 17762932